CLINICAL TRIAL: NCT02597426
Title: A Comprehensive Prospective Cross Sectional Study on the Late Effects of Radical Chemoradiotherapy in Nasopharyngeal Carcinoma Patients Treated in the Intensity-Modulated Radiotherapy Era
Brief Title: Nasopharyngeal Carcinoma Post IMRT
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 15-9063-CE
Record Dates: First submitted 2015-08-18; First posted 2015-11-05 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Intensity-Modulated Radiotherapy; Post treatment
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient: Nasopharyngeal carcinoma (NPC) patients who are disease free more than four years after definitive management with radiotherapy +/- chemotherapy who were treated with Intensity-Modulated Radiotherapy (IMRT), study will involve Collection of demographic data, endocrine assessment (Pituitary and Thyroid), Patient reported outcomes (Quality of Life Questionnaire), neurocognitive assessment (Behavioral rating scale) and audiology assessment (Assessment of hearing)
- Caregiver/Family member: Caregivers for patients who consent to participate. Study will involve Frontal Systems Behavior Scale- FrSBe (behavioral rating scale)

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a type of head and neck cancer. The last three decades of research in head and neck radiation oncology have largely focused on improvements in survival, which have mostly come at the cost of long term toxicity for surviving patients.

This is an observational study that is being done to learn about the long-term symptoms and side effects that survivors of nasopharyngeal cancer may have following radiation treatment. This study will include assessment of patient report outcomes, physician-graded adverse events, neurocognitive assessment and endocrine and hearing testing

DETAILED DESCRIPTION:
This study is designed to provide comprehensive cross sectional information on the late toxicities following radical chemoradiotherapy in nasopharyngeal carcinoma in patients who are disease free with a minimum of four years follow-up and who were treated with contemporary radiotherapy techniques (IMRT). This is an observational cross-sectional study which will aim to define the late effects in this population, investigating both well known toxicities identified from studies using earlier radiotherapy techniques (2D and 3D radiotherapy) as well as toxicities which have not been well defined in the current literature and which may be under-recognized and under treated (pituitary function and neurocognitive outcomes).

This study will assess survivors at a single time point four years after completion of their treatment who are disease free. This comprehensive review will include demographic data, clinical assessment, biochemical assessment of hormonal (pituitary and thyroid) function, patient reported outcomes, and quality of life and neurocognitive questionnaires. This study will attempt to comprehensively review these toxicities in a contemporary patient group with modern radiotherapy techniques in an attempt to bridge the gap between current recommended follow up protocols and the actual challenges faced by long term survivors. Some of these factors will be correlated with radiation doses received by the patient to inform on radiation dose thresholds for appropriate toxicities (hypothalamic-pituitary, thyroid, temporal lobe necrosis, neurocognitive performance). Patients will be offered follow-up, if required with appropriate personnel if appropriate, including neuropsychology, endocrinology and otoloryngology.

ELIGIBILITY:
Inclusion Criteria:

All patients with a previous diagnosis of NPC treated with curative intent who are alive and disease free with a minimum of four years of follow up following completion of treatment

* Received treatment with IMRT
* Age 18 or above, no upper limit
* Ability to comply with the protocol

Exclusion Criteria:

* History of recurrent nasopharyngeal disease
* A history of any physical, psychological or social condition which would impair with the ability of the patient to cooperate in this study
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nasopharyngeal carcinoma (NPC) patients who are disease free more than four years after definitive management with radiotherapy +/- chemotherapy who were treated with Intensity-Modulated Radiotherapy (IMRT)
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-06; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of late toxicities( will be measured using CTCAE v 4.0 criteria) | 1 Year
  • Clinical toxicities will be grade according to Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03), a well known toxicity grading scale from 0 (asymptomatic) to 5 (death).
Serum Biochemical Tests for Endocrine Function (fT4, TSH) | 1 Year
  * A single blood test (at same time as the pituitary assessment) will include free thyroxine (fT4; units pmol/L), Thyroid-Stimulating Hormone (TSH; units mIU/L),
  * Biochemical serum deficiencies in morning testing will be scored individually according to CTCAEv4.03
Quality of Life Questionnaires: Functional Assessment of Cancer Therapy (FACT-G, FACT-HN) | 1 Year
  * Quality of life as measured by Functional Assessment of Cancer Therapy-Head & Neck (FACT-HN) and FACIT-Fatigue ranking individual items from 0= not at all to 4 = very much.
  * An overall score is reported on the sum of individual items. The FACT-HN consists of the FACT-G (which consists of 27 questions from physical, social, emotional and functional domains) and a 12-item specific head and neck module. A maximum score for the FACT-HN of 144 reflects the best possible quality of life.
Quality of Life Questionnaires: Functional Assessment of Chronic Illness Therapy-Fatigue (FACT-Fatigue) | 1 Years
  A 13-item specific questionnaire scored using individual items from 0= not at all to 4 = very much collated for a total score.
Quality of Life Questionnaires: Utilities Assessment (EuroQoL - EQ-5D) | 1 YEAR
  A standardized self-reported utility instrument consisting of 5 discrete, 3-level items, and a visual analog scale
Quality of Life Questionnaires: Symptom Burden of Treatment (MD Anderson Symptom Inventory-Head Neck) | 1 YEAR
  • A patient-reported outcome instrument consisting of 28 items, 19 related to common and severe symptoms experienced by cancer patients and 9 specific to head and neck, rated from 0=not present to 10=as bad as you can imagine
Quality of Life Questionnaires: Assessment of Depression and Anxiety (Hospital and Anxiety Depression Score) | 1 YEAR
  A 14 question item scale (7 Anxiety and 7 depression) score 0-3 (each item is individually written) for individual anxiety and depressions scores from 0-21 with validated cut-off points
Assessment of Frontal Lobe Behavior (Frontal Systems Behaviour Scale) | 1 YEAR
  A validated self-rating scale designed to measure the three frontal systems behavioral syndromes: apathy, disinhibition, and executive dysfunction. A 46-item questionnaire rated pre- and post treatment is scored 1=almost never to 5= almost always. Summary scores are calculated and converted to t-scores.
Cognitive Assessment (Montreal Cognitive Assessment - MoCA) | 1 YEAR
  A short cognitive assessment testing several cognitive domains - visuospatial, naming, memory, attention, language, abstraction, delayed recall and orientation. A maximum score is 30.

SECONDARY OUTCOMES:
Association of Radiation Dose with Temporal Lobe Necrosis | 1 Year
  Dose Volume Histograms (DVHs; quantitative radiation dose data delivered to specific organs) will be calculated from initial radiotherapy plans to review association between dose received by the temporal lobe and risk of temporal lobe necrosis.
Association of Radiation Dose with Hearing Loss | 1 Year
  Dose Volume Histograms (DVHs; quantitative radiation dose data delivered to specific organs) will be calculated from initial radiotherapy plans to review association between dose received by the cochlear and vestibulocochlear nerve and risk of hearing loss
Association of Radiation Dose with Cognitive Impairment | 1 Year
  Dose Volume Histograms (DVHs; quantitative radiation dose data delivered to specific organs) will be calculated from initial radiotherapy plans to review association between dose received by the temporal lobe, brain and hippocampus and risk of neurocognitive impairment.
Association of Radiation Dose with Pituitary Dysfunction | 1 Year
  Dose Volume Histograms (DVHs; quantitative radiation dose data delivered to specific organs) will be calculated from initial radiotherapy plans to review association between dose received by the pituitary and risk of hypopituitarism
Association of Radiation Dose with Hypothyroidism | 1 Year
  Dose Volume Histograms (DVHs; quantitative radiation dose data delivered to specific organs) will be calculated from initial radiotherapy plans to review association between dose received by the thyroid gland and risk of hypothyroidism
Association between dysphagia and quality of life | 1 Year
  Correlation between dysphagia and FACT-HN score and EQ-D5
Association between hearing and quality of life | 1 Year
  Correlation between dysphagia and and FACT-HN score and EQ-D5
Association between hearing and quality of life | 1Year
  Correlation between degree of hearing loss (on audiology) and FACT-HN score and EQ-D5
Association between cranial neuropathy and quality of life | 1Year
  Correlation between degree of cranial neuropathy and FACT-HN score and EQ-D5
Association between neurocognitive score (MoCA) and quality of life | 1 Year
  Correlation between Montreal Cognitive Assessment Score and FACT-HN score and EQ-D5
Association between frontal functioning and quality of life | 1 Year
  Correlation between FrSBE (Frontal Systems Behaviour) and FACT-HN score and EQ-D5
Association between pituitary function and quality of life | 1 Year
  Correlation between pituitary function and FACT-HN score and EQ-D5
Association between thyroid function and quality of life | 1 Year
  Correlation between thyrrhoid function and FACT-HN score and EQ-D5

CONTACTS AND LOCATIONS:
Overall Officials: John N Waldron, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada